CLINICAL TRIAL: NCT01505894
Title: Safety, Tolerability Pharmacokinetics and Pharmacodynamics of Multiple Rising Doses of BI 409306 Film-coated Tablets Given Orally q.d. or Bid for 14 Days in Young Healthy and Elderly Healthy Male/Female Volunteers (Randomised, Double-blind, Placebo Controlled Within Dose Groups Phase I Study)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.2; 2011-002369-39 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306

ARMS (9):
- Placebo - Young Subjects (Placebo Comparator): Placebo - Young Subjects
  Interventions: Drug: Placebo
- Placebo - Elderly Subjects (Placebo Comparator): Placebo - Elderly Subjects
  Interventions: Drug: Placebo
- BI 409306 25 mg - Young Subjects QD (Experimental): 25 milligram (mg) of BI 409306 were administered in young subjects once daily (QD).
  Interventions: Drug: BI 409306
- BI 409306 25 mg - Elderly Subjects QD (Experimental): 25 mg of BI 409306 were administered in elderly subjects once daily (QD).
  Interventions: Drug: BI 409306
- BI 409306 50 mg - Young Subjects QD (Experimental): 50 mg of BI 409306 were administered in young subjects once daily (QD).
  Interventions: Drug: BI 409306
- BI 409306 50 mg - Young Subjects BID (Experimental): 50 mg of BI 409306 were administered in young subjects twice daily (BID).
  Interventions: Drug: BI 409306
- BI 409306 50 mg - Elderly Subjects QD (Experimental): 50 mg of BI 409306 were administered in elderly subjects once daily
  Interventions: Drug: BI 409306
- BI 409306 100 mg - Young Subjects QD (Experimental): 100 mg of BI 409306 were administered in young subjects once daily (QD).
  Interventions: Drug: BI 409306
- BI 409306 100 mg - Elderly Subjects QD (Experimental): 100 mg of BI 409306 were administered in elderly subjects once daily (QD).
  Interventions: Drug: BI 409306

INTERVENTIONS:
Drug: BI 409306 — Film-coated tablet
  Arms: BI 409306 100 mg - Elderly Subjects QD; BI 409306 100 mg - Young Subjects QD; BI 409306 25 mg - Elderly Subjects QD; BI 409306 25 mg - Young Subjects QD; BI 409306 50 mg - Elderly Subjects QD; BI 409306 50 mg - Young Subjects BID; BI 409306 50 mg - Young Subjects QD
Drug: Placebo — Film-coated tablet
  Arms: Placebo - Elderly Subjects; Placebo - Young Subjects

SUMMARY:
The primary objective of this trial was to investigate safety and tolerability of multiple doses of BI 409306 in healthy young and elderly volunteers.

The secondary objective was to explore the pharmacokinetics and pharmacodynamics of multiple doses of BI 409306 in healthy young and elderly volunteers

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age >21 and Age <50 years for young healthy volunteers or Age >65 and Age <80 years for elderly healthy volunteers
3. BMI >18.5 and BMI <29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.
5. For female subjects: Female subjects must be surgically sterilized or postmenopausal. Surgical sterilization or hysterectomy must have occurred at least 6 months prior to screening. Menopausal women must have no regular menstrual bleeding for at least 2 years prior to screening.

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (including but not limited to any kind of seizures, stroke or psychiatric disorders)
6. History or evidence of relevant orthostatic reaction (drop in systolic blood pressure (SBP) >20 mm Hg and increase in heart rate > 30 bpm after 2 minutes standing relative to supine data), fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of any drugs within 14 days or drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within four weeks prior to administration or during the trial
12. Smoker (> 5 cigarettes or > 1 cigars or > 1 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 20 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance in the judgment of investigator
19. Inability to comply with dietary regimen of trial site
20. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc F interval >430 ms in males and >450 ms in females);
21. A history of additional risk factors for Torsades de points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.2.1 Boehringer Ingelheim Investigational Site, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is randomised, placebo control, double blind, phase 1, pharmacokinetic study in healthy young and elderly subjects.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended a specialist sites which ensured that they met all of the inclusion and none of exclusion criteria. Participants were not to be entered to trial treatment if any one of the specific entry criteria was violated.
Groups:
- Placebo- Young Subjects: Healthy young subjects administered with placebo (matching BI409306) orally once daily for 14 days or twice daily on Days 2 to 13 with two single doses on the Days 1 and 14 for dose group 2.
- Placebo-Elderly Subjects Once Daily (QD): Healthy elderly subjects administered with placebo (matching BI409306) orally once daily (QD) for 14 days.
- BI 409306 25 Milligram- Young Subjects (QD): Healthy young subjects administered with BI 409306 25 milligram film coated tablet orally once daily for 14 days.
- BI 409306 25 Milligram- Elderly Subjects (QD): Healthy elderly subjects administered with BI 409306 25 milligram film coated tablet orally once daily for 14 days.
- BI 409306 50 Milligram- Young Subjects (QD): Healthy young subjects administered with BI 409306 50 milligram film coated tablet orally once daily for 14 days.
- BI 409306 50 Milligram- Young Subjects (BID): Healthy young subjects administered with BI 409306 50 milligram film coated tablet orally twice daily (BID) from day 2 to 13 , and once daily on days 1 and 14. (Dose group 2).
- BI 409306 50 Milligram- Elderly Subjects (QD): Healthy elderly subjects administered with BI 409306 50 milligram film coated tablet orally once daily for 14 days.
- BI 409306 100 Milligram- Young Subjects (QD): Healthy young subjects administered with BI 409306 100 milligram film coated tablet orally once daily for 14 days.
- BI 409306 100 Milligram- Elderly Subjects (QD): Healthy elderly subjects administered with BI 409306 100 milligram film coated tablet orally once daily for 14 days.
Period: Overall Study
Arm/Group | Placebo- Young Subjects | Placebo-Elderly Subjects Once Daily (QD) | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Started | 12 | 9 | 9 | 9 | 9 | 9 | 8 | 9 | 9
Completed | 11 | 9 | 9 | 9 | 8 | 9 | 8 | 9 | 9
Not Completed | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other than specified | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: Included all subjects who are treated with BI 409306.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo- Young Subjects | Placebo-Elderly Subjects Once Daily (QD) | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD) | Total
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 9 | 8 | 9 | 9 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years off all subjects in the study Population: Treated Set: Included all subjects who are treated with BI 409306.
  Years
    Young Subjects: number analyzed (Participants) | 12 | 0 | 9 | 0 | 9 | 9 | 0 | 9 | 0 | 48
    Young Subjects | 41.8 (9.7) |  | 42.2 (6.6) |  | 42.1 (8.1) | 41.9 (7.9) |  | 42.2 (6.3) |  | 42.0 (7.6)
    Elderly Subjects: number analyzed (Participants) | 0 | 9 | 0 | 9 | 0 | 0 | 8 | 0 | 9 | 35
    Elderly Subjects |  | 67.6 (3.0) |  | 69.1 (3.1) |  |  | 70.5 (4.0) |  | 67.9 (3.6) | 68.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution of all subjects in the study Population: Treated Set: Included all subjects who are treated with BI 409306.
  Participants
    Female | 4 | 7 | 2 | 5 | 4 | 3 | 6 | 2 | 3 | 36
    Male | 8 | 2 | 7 | 4 | 5 | 6 | 2 | 7 | 6 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of all included subjects in the study. Ethnicity data was not collected for this trial. Population: Treated Set: Included all subjects who are treated with BI 409306.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 12 | 9 | 9 | 9 | 8 | 9 | 8 | 9 | 9 | 82
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Maximum Concentration of BI 409306 in Plasma (Cmax)
Description: Maximum measured concentration of the BI 409306 in plasma after first dose.
Time Frame: On day 1, at -2:00 hours (pre dose) and at 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 hours after the first dose.
Population: Pharmacokinetic Analysis Set (PKS): Included all subjects in the treated set who provided at least 1 evaluable observation for a pharmacokinetic endpoint in at least 1 treatment period (single dose or multiple dose segment) and had no important protocol violation relevant to the evaluation of pharmacokinetics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles/Litre (nmol/L)
Arm/Group | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 8 | 9 | 9
Nanomoles/Litre (nmol/L) | 245 (130) | 376 (48.0) | 565 (84.6) | 696 (47.8) | 1100 (58.5) | 1030 (79.2) | 1840 (68.1)

2. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of BI 409306 in Plasma (Tmax)
Description: Time from dosing to maximum measured concentration of BI 409306 in plasma (Tmax) after the first dose.
Time Frame: On day 1, at -2:00 hours (pre-dose) and at 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 hours after the first dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 8 | 9 | 9
Hour (h) | 0.750 [0.500 to 1.52] | 0.500 [0.167 to 0.750] | 0.500 [0.333 to 0.750] | 0.750 [0.333 to 0.750] | 0.333 [0.167 to 1.00] | 0.500 [0.333 to 0.750] | 0.500 [0.333 to 1.50]

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 extrapolated to infinity after first dose.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole*Hour/Litre (nmol*h/L)
Arm/Group | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 8 | 9 | 9
Nanomole*Hour/Litre (nmol*h/L) | 548 (142) | 594 (48.6) | 955 (97.6) | 1140 (54.0) | 1510 (70.5) | 1620 (60.1) | 2840 (56.1)

4. Secondary Outcome: Maximum Concentration of BI 409306 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: Maximum measured concentration of the BI 409306 in plasma at steady state over a uniform dosing interval τ after last dose.
Time Frame: At 312:00 hours (pre dose) and at 312:10 , 312:20, 312:30, 312:45, 313:00, 313:30, 314:00, 314:30, 315:00, 316:00, 318:00, 320:00, 322:00, 324:00, 326:00, 336:00, 360:00, 384:00 hours post dose, for once daily and twice daily treatment.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole/Litre (nmol/L)
Arm/Group | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 8 | 9 | 9
Nanomole/Litre (nmol/L) | 348 (71.4) | 444 (44.2) | 663 (98.0) | 596 (42.8) | 1250 (76.6) | 1260 (55.4) | 2150 (87.0)

5. Secondary Outcome: Time to Achieve Maximum Concentration of BI 409306 in Plasma at Steady State (Tmax,ss)
Description: Time from last dosing until the maximum concentration of the analyte in plasma is reached at steady state after last dose on day 14.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 8 | 9 | 9
Hour (h) | 0.750 [0.333 to 0.783] | 0.500 [0.333 to 0.750] | 0.625 [0.333 to 1.02] | 0.750 [0.500 to 1.00] | 0.417 [0.167 to 1.50] | 0.500 [0.333 to 0.750] | 0.333 [0.167 to 1.50]

6. Secondary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma at Steady State (AUCτ,ss)
Description: This endpoint calculates area under the concentration-time curve of BI 409306 in plasma at steady state over a uniform dosing interval τ after last dose on day 14.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole*Hour/Litre (nmol*h/L)
Arm/Group | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 8 | 9 | 9
Nanomole*Hour/Litre (nmol*h/L) | 747 (93.1) | 621 (55.8) | 1070 (125) | 1100 (52.4) | 1710 (83.6) | 1960 (64.3) | 3990 (119)

7. Primary Outcome: Number of Young and Elderly Subjects With On-treatment Adverse Events by Treatment Group
Description: An adverse event is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a subject in a clinical investigation who received a pharmaceutical product.
Time Frame: From first drug administration until the end-of-trial examination, up to 28 days.
Population: Treated Set (TS): Included all subjects who are treated with BI 409306.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Young Subjects | Placebo-Elderly Subjects Once Daily (QD) | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 9 | 8 | 9 | 9
Participants | 6 | 3 | 5 | 6 | 4 | 8 | 5 | 8 | 8

8. Primary Outcome: Number of Participants With Clinically Relevant Abnormal Findings in Vital Signs, 12-lead ECG, Clinical Laboratory Tests, Physical Examination, Ophthalmological Examination and Suicidality Assessment
Description: Number of participants with clinically relevant abnormal findings, as judged by investigator and reported as adverse event (AE), in vital signs (blood pressure, pulse rate, orthostatic test), 12-lead electrocardiogram (ECG), clinical laboratory tests (haematology, clinical chemistry, urinalysis) , physical examination, ophthalmological examination and suicidality assessment.
Time Frame: From first drug administration until the end-of-trial examination, up to 28 days.
Population: Treated Set (TS): Included all subjects who are treated with BI 409306.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Young Subjects | Placebo-Elderly Subjects Once Daily (QD) | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 9 | 8 | 9 | 9
Participants
  Vital signs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  12-lead ECG | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clinical laboratory test | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Physical examiniation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ophthalmological examination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Suicidality assessment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants Per Category of Global Tolerability Assessed by the Investigator
Description: The investigator assessed tolerability based on adverse events and the laboratory evaluation and classified the overall tolerability according to the categories 'good', 'satisfactory', 'not satisfactory', and 'bad'. Investigator judgement based on clinical findings: "good" - No or mild adverse events (AEs) and no clinically significant (NCS) findings in any clinical assessments; "satisfactory" - mild or moderate AEs, NCS clinical findings; "not satisfactory" - moderate/severe AEs and/or clinically significant (CS) findings.
Time Frame: From first drug administration until the end-of-trial examination, up to 28 days.
Population: Treated Set (TS): Included all subjects who are treated with BI 409306.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Young Subjects | Placebo-Elderly Subjects Once Daily (QD) | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 9 | 8 | 9 | 9
Participants
  Good | 11 | 9 | 9 | 9 | 9 | 9 | 8 | 9 | 8
  Satisfactory | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not satisfactory | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bad | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not assessable | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Abnormal Findings in Color Discrimination Test
Description: Color vision was tested using the Ishihara test for color deficiency. The test consisted of a number of plates, called Ishihara plates, each of which contains a circle of dots of differing color and size. Within the pattern some dots form a number visible to those with normal color vision and invisible, or difficult to see, for those with a color vision deficiency. Participants with abnormal findings in color discrimination test are participants, who are not able to recognize the sign on the presented table.
Time Frame: From first drug administration until the end-of-trial examination, up to 28 days.
Population: Treated Set (TS): Included all subjects who are treated with BI 409306.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Young Subjects | Placebo-Elderly Subjects Once Daily (QD) | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 9 | 8 | 9 | 9
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Abnormal Findings in Visual Acuity Test
Description: Snellen chart was used to measure visual acuity. It measures the smallest line that a participant was able to read at a distance of 3 meter. Participants with abnormal findings in visual acuity test are participants, who are not able to recognize the letters on the line 3.
Time Frame: From first drug administration until the end-of-trial examination, up to 28 days.
Population: Treated Set (TS): Included all subjects who are treated with BI 409306.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Young Subjects | Placebo-Elderly Subjects Once Daily (QD) | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 9 | 8 | 9 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first drug administration until the end-of-trial examination, up to 28 days.
Description: Treated set was used for analysis of adverse events data.
Arm/Group | Placebo- Young Subjects | Placebo-Elderly Subjects Once Daily (QD) | BI 409306 25 Milligram- Young Subjects (QD) | BI 409306 25 Milligram- Elderly Subjects (QD) | BI 409306 50 Milligram- Young Subjects (QD) | BI 409306 50 Milligram- Young Subjects (BID) | BI 409306 50 Milligram- Elderly Subjects (QD) | BI 409306 100 Milligram- Young Subjects (QD) | BI 409306 100 Milligram- Elderly Subjects (QD)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 6/12 | 3/9 | 5/9 | 6/9 | 4/9 | 8/9 | 5/8 | 8/9 | 8/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo- Young Subjects (N=12) | Placebo-Elderly Subjects Once Daily (QD) (N=9) | BI 409306 25 Milligram- Young Subjects (QD) (N=9) | BI 409306 25 Milligram- Elderly Subjects (QD) (N=9) | BI 409306 50 Milligram- Young Subjects (QD) (N=9) | BI 409306 50 Milligram- Young Subjects (BID) (N=9) | BI 409306 50 Milligram- Elderly Subjects (QD) (N=8) | BI 409306 100 Milligram- Young Subjects (QD) (N=9) | BI 409306 100 Milligram- Elderly Subjects (QD) (N=9)
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 5 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 5
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Visual impairment (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 0 | 2 | 3 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.